CLINICAL TRIAL: NCT05178823
Title: Short- and Long Term Antibacterial Effects of a Single Rinse With Different Mouthwashes: a Randomized Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Solumium
Record Dates: First submitted 2021-12-17; First posted 2022-01-05 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Gingival Diseases; Caries
Keywords: single rinse; mouthwash; chlorine dioxide; S. mutans
MeSH Terms: conditions — Gingival Diseases | interventions — chlorine dioxide; Oils, Volatile; Sodium Fluoride; zinc chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Corsodyl (Active Comparator): Chlorhexidine
  Interventions: Drug: Chlorhexidine mouthwash
- Solumium Oral (Experimental): Chlorine dioxide
  Interventions: Drug: Chlorhexidine mouthwash
- Listerine Total Care (Experimental): Essential oils, sodium fluoride, zinc chloride
  Interventions: Drug: Chlorhexidine mouthwash
- BioGate Si*CLEAN (Experimental): Microsilver
  Interventions: Drug: Chlorhexidine mouthwash

INTERVENTIONS:
Drug: Chlorhexidine mouthwash — Comparison of oral rinses
  Other Names: chlorine dioxide; essential oils, sodium fluoride, zinc chloride; microsilver

SUMMARY:
Objectives: To reduce the microbial level in the aerosol created during dental procedures is essential in avoiding infections. The aim of this study was to examine the change of Streptococcus mutans (S. mutans) and the total bacterial load in human saliva in vivo after a single rinse with different mouthwashes.

Material and methods: One mL unstimulated saliva was collected from volunteers with poor oral hygiene at baseline and 5 min after a one-min rinsing with Solumium Oral® (hyper-pure 0.0015% chlorine dioxide; ClO2), Listerine Total Care®, Corsodyl® (0.2% chlorhexidine-digluconate; CHX), or BioGate Si*CLEAN for bacterial investigation. In a second study volunteers rinsed with 0.003% ClO2 or CHX for one-min and saliva was collected at baseline, after 5 and 90 min. After plating the total plate and S. mutans colony numbers were determined.

DETAILED DESCRIPTION:
Sample and procedure In the first study we collected 1 mL of unstimulated whole saliva by spitting participants into a sterile Eppendorf tube at baseline and 5 min after rinsing with 5 mL of 4 different types of commercially available mouthwashes from identical opaque-coded flasks. From our clinical ambulance randomly selected 145 patients assessed for eligibility. Inclusion criteria were: DMF≥10, minimum 5 active caries and PSR≥2. Exclusion criteria were: smoking, a history of antibiotic, or probiotic use 3 months prior to sampling, or known allergy to any of the ingredients of mouthwashes being tested. Twenty five patients were excluded (19 of these based on the criteria above and 6 refused to participate). One hundred and twenty volunteering patients (42±8 years) with poor oral hygiene were selected to participate in the study. All eligible subjects were given oral and written information about the products and the purpose of the study and were asked to sign an informed consent form. Volunteers were randomly assigned to the tests and the positive control (Corsodyl®) groups. Randomization was performed using computer-generated random numbers. The randomization and the allocation of rinse aids were carried out by a person not directly involved in the research project. The volunteers rinsed for 1 min, with a 20-fold dilution of hyper-pure 0.03 % ClO2 (Solumium Oral®, final concentration: 0.0015%), Corsodyl® (0.2% CHX), Listerine Total Care® (essential oils, sodium fluoride, zinc chloride), or BioGate Si*CLEAN® (microsilver) (30 individuals in each mouthwash group).

In the second study randomly chosen 26 medical student volunteers (20±3 years) rinsed with 5 mL of 10-fold diluted hyper-pure ClO2 (final concentration: 0.003%) or Corsodyl® for 1 min, and their unstimulated whole saliva was collected as above at base line and after 5 and 90 minutes (13 individuals in each mouthwash group). The restrictions on the oral hygiene of the volunteers were: DMF≥5, minimum 1 active caries, PSR≥1 and exclusion categories were the same as in the first study. The management of eligible subjects, their randomization and the allocation of rinse aids in same opaque-coded flasks were also exactly identical to the first study. Eleven volunteers were excluded from this study (9 of these based on the criteria above and 2 refused to participate).

The saliva samples were stored in Eppendorf tubes used for collection at air-conditioned room temperature and processed within two hours. A dilution series was prepared from the samples in physiological salt solution. To determine our pre-specified primary outcome, the total bacterial count and the S. mutans number (CFU/ml) blood and Mitis-Salivarius (Difco, Becton-Dickinson, Hungary) agars were inoculated, respectively. Cultivation was carried out at 37 °C, 5 % CO2 and took 2 days. The CFU counting researcher did not know which plates were exposed to each treatment.

ELIGIBILITY:
Inclusion Criteria:

* DMF≥10,
* minimum 5 active caries
* PSR≥2

Exclusion Criteria:

* smoking,
* a history of antibiotic, or probiotic use 3 months prior to sampling
* known allergy to any of the ingredients of mouthwashes being tested

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Salivary bacterial CFU/mL | 1 or 90 min after rinsing
  Salivary bacterial CFU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Zsolt Lohinai, PHD, Principal Investigator — Semmelweis University, Department of Conservative Dentistry
Locations (1):
- Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Herczegh A, Gyurkovics M, Agababyan H, Ghidan A, Lohinai Z. Comparing the efficacy of hyper-pure chlorine-dioxide with other oral antiseptics on oral pathogen microorganisms and biofilm in vitro. Acta Microbiol Immunol Hung. 2013 Sep;60(3):359-73. doi: 10.1556/AMicr.60.2013.3.10. PMID 24060558